CLINICAL TRIAL: NCT00000289
Title: Role of Metabolites in Nicotine Dependence (3)
Brief Title: Role of Metabolites in Nicotine Dependence (3) - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-6; P50-09259-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-12

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Ondansetron

INTERVENTIONS:
Drug: Ondansetron

SUMMARY:
The purpose of this study is to determine the effects of various doses of ondansetron transdermal nicotine replacement on tobacco withdrawal symptoms.

DETAILED DESCRIPTION:
Previous studies have shown that cotinine, a metabolite of nicotine, antagonizes the beneficial effects of the nicotine patch in redugin withdrawal symptoms. Studies have also shown that cotinine enhances serotonin levels. This study examined the effects of several doses of a 5HT3 antagonist, ondanstron, in combination with the nicotine patch. This medication has been observed to reduce nicotine withdrawal symptoms in rats. These effects were compared to the nicotine patch alone. The results of this study produced some modest effects showing that the 8mg dose of ondansetron suppressed tobacco withdrawal symptoms to a greater extent than the nicotine patch alone.

ELIGIBILITY:
Inclusion Criteria:

Male/Female subjects ages 21-45 years inclusive, with a smoking history of at least 15 cigarettes daily (greater than or equal to 50) for at least 1 yr. Subject is in good health as verified by medical history, screening examination, and screening laboratory tests as outlined above. Subject has provided written informed consent to participate in the study and is motivated to stop smoking. Subject has experienced at least 4 withdrawal symptoms upon abstinence.

Exclusion Criteria:

History of myocardial infarction, angina pectoris, sustained or episodic cardiac arrhythmias, symptomatic peripheral vascular disease, current peptic ulcer disease or any other medical condition which the physician investigator deems inappropriate for subject participation. Insulin-dependent diabetes. Pregnant or lactating, or not using adequate birth control methods. Requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history (less than 1yr). Chronic use of systemic steroids or antihistamines. Abuse of alcohol or any other recreational or prescription drug (more than 3 drinks per day or 21 drinks per wk). use of any other nicotine products, including smokeless tobacco, cigars and nicotine replacement products. Inability to fulfill all scheduled visits and examination procedures throughout the study period. History of schizophrenia or manic depressive disorder. Recent history of other psychiatric illness (less than 1yr since last episode of major depressive episode).

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1998-05; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective effects
Physiological effects
Performance effects

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States